CLINICAL TRIAL: NCT01478724
Title: Effects of Proteins Fraction Derived From Milk on Bone Mineral Density and Bone Metabolism in Healthy Postmenopausal Women
Brief Title: Effects of Proteins Fraction Derived From Milk on Osteoporosis Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soredab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SORBONE
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Animal proteins
  Interventions: Dietary Supplement: Milk proteins fraction
- Milk protein fraction dose 1 (Experimental)
  Interventions: Dietary Supplement: Milk proteins fraction
- Milk protein fraction dose 2 (Experimental)
  Interventions: Dietary Supplement: Milk proteins fraction

INTERVENTIONS:
Dietary Supplement: Milk proteins fraction — capsules, one per day, 24 months

SUMMARY:
Osteoporosis is defined as a systemic skeletal disease characterised by low bone mass and microarchitectural deterioration of bone tissue, with a consequent increase in bone fragility and susceptibility to fracture. Osteoporosis is a serious public health problem that is responsible for approximately 3 million women with osteoporosis in France, with approximately 150,000 cases per year occurring in vertebral fractures, of which only one third would be diagnosed and 50,000 hip fractures (causing death in 20% of cases). The frequency of the disease increases with age, particularly among women: 10% among women aged 60 years and 20% among women aged 65 and 40% among women aged 75. At menopause, oestrogen deficiency causes alterations of the immune system, decreased bone formation, microarchitectural deterioration and a decrease in bone mass. Various factors may contribute to this decrease in bone density such as diet, lifestyle, or the genetic background.

According to prospective studies, an overexpression of 135% of hip fractures is expected at European level in 50 years. Therefore, it is interesting to develop new prevention approaches aimed at maintaining the healthy aging population. Nutritional researches can consider setting up a real prevention.

Studies suggest that specific milk protein fraction contain factors able to promote bone formation, inhibit bone resorption in vitro. In animal model, they showed that the specific fraction prevents bone loss in aged ovariectomised rats by reducing bone resorption. Furthermore, in human volunteers, a supplementation with the specific milk protein fraction maintains balanced bone remodelling and increase bone mineral density. For example, in healthy postmenopausal women, it has been reported that a mean rate of gain of lumbar BMD in the MPF group (1.21%) was significantly higher than in placebo group (-0.66%; p<0.05).

The objective of this study is to assess the efficacy of daily consumption of the milk proteins fraction on bone mineral density improvement in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian Female
* Natural or surgical menopause between 1 and 5 years
* Aged between 50 to 65 years
* BMI between 19 and 30 kg/m²

Exclusion Criteria:

* Medications: oral steroidal anti-inflammatory, anti-osteoporotic treatment, hormone replacement therapy
* Low bone mineral density (T-score<-3
* Diseases affecting bone metabolism(Paget's disease, Cushing's disease, thyroid disease...)
* Intolerance or allergy to milk proteins and allergy to soy or soy lecithin
* Heavy smoking
* Excessive alcohol drinking
* Intensive sports practice according to the investigator

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
lumbar spine bone mineral density | 24 months

SECONDARY OUTCOMES:
femoral bone mineral density | 12 and 24 months
lumbar spine bone mineral density | 12 months
bone remodelling biomarkers | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Roux, PUPH, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin hospital, Paris, France